CLINICAL TRIAL: NCT00844272
Title: Psychoeducation Reaches HCV-infected Methadone/Buprenorphine Substituted Patients in Standard Antiviral Treatment
Acronym: Permit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Prof. Dr. med. Jens Reimer, Director Centre for Interdisciplinäry Addiction Research, Universitätsklinikum Hamburg-Eppendorf
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIAR-PERMIT
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Intravenous Drug Abuse; Chronic Hepatitis C
Keywords: Opiate Dependence; Chronic Hepatitis C
MeSH Terms: conditions — Substance Abuse, Intravenous; Hepatitis C, Chronic; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychoeducation (Experimental): PE group sessions lasted 60 minutes and were carried out under continuous supervision. The manualised program was especially tailored to (former) IDUs in HCV treatment, containing the following aspects:
  * Module 1: HCV infection and symptoms, course of illness, interaction with opioid dependence, further problems and risk factors
  * Module 2: HCV treatment, side effects, psychiatric and somatic comorbidities, reinfection and drug use, risk behaviour
  * Module 3: Coping strategies, resources and self-help, effective use of health-care support, the role of social environment, healthy living & nutrition
  Interventions: Behavioral: Psychoeducation
- Treatment as usual (No Intervention): Control group did not received no intervention.

INTERVENTIONS:
Behavioral: Psychoeducation — Group-therapeutic intervention with 12 sessions plus 5 update sessions with 24-week therapy duration and/or 12 sessions plus 10 update sessions with 48-week therapy duration Module I: Create understanding, resources, problems and solutions Module II: Information on hepatitis C infection Module III: Information on treatment Module IV: Specific information on depression and withdrawal symptoms under interferon The meetings take a minimum of 60 min. time, should be once weekly. The group size should lie between 6 and 12 participants.
  The group leaders are trained in performance of the psycho-education.
  Arms: Psychoeducation

SUMMARY:
Study objective: Feasibility and efficacy of a standardised psychosocial intervention (psychoeducation) in substituted opioid dependent patients

DETAILED DESCRIPTION:
Primary objective:

* Retention in antiviral treatment (feasibility)

Secondary objectives:

* Mental Health Mental health is monitored by means of the Symptom Checklist 90-R (SCL-90-R). Its sum score, the Global Severity Index (GSI), serves as indicator. Mental health will be regarded as stable in case of a change of less than 6 GSI-points, otherwise mental health will be regarded as improved (GSI - 6 points) or decreased (GSI + 6 points).
* Course of Addiction Course of addiction under antiviral treatment will be monitored according to retention in substitution treatment, compliance with scheduled visits, and co-consumption of illicit drugs (patients record, urinalysis).
* Sustained viral response (SVR) SVR as measured by polymerase chain reaction 6 months after per protocol antiviral treatment (ITT-analysis).

ELIGIBILITY:
Inclusion Criteria:

* Women and men at the age of 18 to 70 years
* Opiate dependence according to ICD-10
* Stable substitution (i.e. either keeping the last 5 dates or fulfilling criteria for the Take Home assignment)
* Proof of HCV by means of PCR
* Patient must be therapy naive regarding the hepatitis C (no preceding treatment attempts with interferon and/or Ribavirin)
* Ability to comprehend und follow the study protocol
* Compensated liver disease with the following haematological and biochemical minimum criteria:

  1. Leukocytes ≥ 3.000/mm3
  2. Neutrophile granulocytes ≥ 1.500/mm3
  3. Thrombocytes ≥ 90.000/mm3
  4. Direct and indirect bilirubin within the standard range (if not factors, which are not hepatitis-conditioned, as M. Meulengracht, represent an explanation for the increase of the indirect bilirubin; in these cases the indirect bilirubin must be less than 3.0 mg/dl or 51.3 µmol/l)
  5. Albumin within the standard range
  6. Creatinine within the standard range
* TSH (Thyreotropine) within the standard range of the test laboratory
* Normal blood sugar value for non-diabetics or haemoglobin A1c max. 8.5% for diabetics (induced by pharmacotherapy and/or diet controls). An eye examination is required in diabetics.
* Haemoglobin values ≥ 12 mg/dl for women and/or ≥ 13 mg/dl for men
* ANA ≤ 1:160
* In patients with cirrhosis or transition to cirrhosis: exclusion of hepatocellular carcinoma
* Readiness to abstain from alcohol during interferon treatment.
* Negative pregnancy test in female patients within 24 hours before the first dose
* Regular confirmation that sexual active women at the age capable of child-bearing and/or sexual active men use two reliable methods of contraception during interferon / ribavirin treatment and six months thereafter, one contraception method with barrier effect (e.g. condom, diaphragm)
* Female patients may not breastfeed during interferon / ribavirin treatment.

Exclusion Criteria:

* Decompensated liver cirrhosis (Child-Pugh B or C)
* Haemochromatosis
* Lack of Alfa-1-Antitrypsin (homozygote - PIZZ)
* Morbus-Wilson
* positive proof of HBsAg, anti- HIV or anti- HAV IgM antibodies
* Autoimmune diseases (e.g. autoimmune hepatitis, autoimmune thyroid disease, rheumatoid arthritis)
* Kidney failure (Creatinine > 1,5 mg/dl)
* Liver- or kidney-transplantation
* Hyperlipidemia (Cholesterol > 1,5-times above the upper standard value)
* Clinically manifested gout
* Severe heart insufficiency
* Severe coronary heart disease
* Patients with cardiac pacemaker
* Severe chronic pulmonary diseases (e.g. COPD)
* Serious psychological illness, in particular severe depression
* Epilepsy
* Oesophagus varicose in the prehistory
* Patient with high anaemia risk (e.g. Thalassaemia)
* Retinopathy
* Severe other illness
* Patients, who cannot follow the study conditions
* Male partners of pregnant women
* Current desire to have children / no safe contraception under therapy and until including 6 months after study end
* Participation in a clinical study within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2005-05; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Retention in antiviral treatment (feasibility) | within the first 24/48 weeks

SECONDARY OUTCOMES:
Psychological health | within the first 24/48 weeks
Medical process on the basis of retention in substitution treatment | within the first 24/48 weeks
Permanent virus suppression | within the first 24/48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Gölz, MD, Principal Investigator — Praxiszentrum Kaiserdamm

REFERENCES:
- [Derived] Reimer J, Schmidt CS, Schulte B, Gansefort D, Golz J, Gerken G, Scherbaum N, Verthein U, Backmund M. Psychoeducation improves hepatitis C virus treatment during opioid substitution therapy: a controlled, prospective multicenter trial. Clin Infect Dis. 2013 Aug;57 Suppl 2:S97-104. doi: 10.1093/cid/cit307. PMID 23884073